CLINICAL TRIAL: NCT04103307
Title: Improving Outcomes in Patients Receiving Continuous Renal Replacement Therapy for Acute Kidney Injury by Cooling Blood in the Dialysis Circuit (CRRiTiCool): a Randomized Controlled Trial
Brief Title: Continuous Renal Replacement Therapy for Acute Kidney Injury by Cooling Blood
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment was not feasible due to COVID-19 pandemic so study was stopped
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Marat Slessarev, Assistant Professor of Medicine, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113951
Record Dates: First submitted 2019-08-09; First posted 2019-09-25 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury; Continuous Renal Replacement Therapy
Keywords: Cooling; CRRT
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: The participants will receive CRRT in the form of CVVH or CVVHDF using the PrisMaxTM dialysis machine (Baxter Healthcare Corporation) according to local standard operating procedures. Filter anticoagulation will be maintained using either no anticoagulation, regional citrate or heparin. The TherMax™ blood warmer will be used when required to maintain a minimum body temperature.
  All participants will undergo CRRT via a temporary double-lumen hemodialysis catheter inserted into a central vein (internal jugular vein, subclavian vein, femoral vein).
  The standard of care entails continuous dialysis therapy for as long as deemed clinically necessary by the doctor. An external heater is used to rewarm the blood before delivering it back to the patient. If assigned to the intervention group, cool blood will be received during continuous dialysis. The cool blood will be delivered by having the heater set to 35.5°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Standard of care (No Intervention): Participants in the control group will receive standard-of-care CRRT prescriptions, and have the returning venous blood warmed with an external blood warmer to a temperature of 37°C. The blood warmer temperature will be adjusted by the CRRT nurse as per usual practice to maintain normothermia.
- Intervention: Cooling (Experimental): Participants in the intervention group will receive standard of care CRRT prescriptions and have the blood warmer set to 35.5°C, as long as the nasopharyngeal temperature remains above 35.5°C.
  Interventions: Procedure: Dialysis cooling

INTERVENTIONS:
Procedure: Dialysis cooling — Cooling the blood in the CRRT circuit during delivery
  Arms: Intervention: Cooling

SUMMARY:
Acute kidney injury (AKI) is common in intensive care unit (ICU) patients and is associated with longer hospital stays and worse survival. The mortality rate of critically ill patients in the ICU who receive renal replacement therapy for AKI ranges between 50-80%, cardiovascular disease being the second largest cause of death. A previous pilot study from the investigator's group showed that myocardial stunning occurs in AKI patients during continuous renal replacement therapy (CRRT) and may explain the high cardiovascular mortality in this population. In the chronic intermittent dialysis setting, mild dialysate cooling was shown to improve intradialytic hemodynamic stability and prevent myocardial stunning. The aim of this study is to find out whether cooling the blood in the CRRT circuit is an effective intervention to prevent myocardial stunning in AKI patients undergoing CRRT and improve patient outcomes.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized, open label, controlled trial comparing standard-of-care temperature management with blood cooling CRRT. We will recruit approximately 140 patients (70 in each group) from the Medical Surgical Intensive Care Unit at University Hospital and The Critical Care Trauma Center at Victoria Hospital in London, Ontario.

The study team will randomize patients with acute kidney injury requiring continuous dialysis therapy into one of two groups; either to standard of care continuous dialysis therapy or to cool blood continuous dialysis therapy. All therapy will be delivered using the Baxter PrisMaxTM CRRT machine with TherMaxTM blood warmer.

All participants will undergo a series of echocardiograms (ultrasound of your heart) prior to continuous dialysis therapy initiation, 4-12 hours into therapy, for up to 7 days after therapy initiation, and at discharge from the intensive care unit. Blood work will be collected at 4 time points, prior to continuous dialysis therapy initiation, 4-12 hours into therapy, 24 hours into therapy, and at ICU discharge.

Hourly nasopharyngeal and skin temperatures will be collected. Oral temperature will be collected every four hours.

ELIGIBILITY:
Inclusion Criteria:

* AKI as defined by 2012 AKI KDIGO guidelines requiring CRRT.
* Patient's core temperature between 35°C and 40°C at the time of recruitment.
* Age 18 years old and older.

Exclusion Criteria:

* Hypothermia (patient core temperature <35°C) at the time of recruitment
* Extreme hyperthermia or hyperpyrexia (patient core temperature >40°C) at the time of recruitment.
* Contraindication to cooling (e.g., hemorrhagic shock or severe coagulopathy)
* Patients undergoing targeted temperature management for cardiac arrest.
* Chronic kidney disease stage 5 as defined by CKD KDIGO guidelines [19] requiring renal replacement therapy prior to recruitment.
* Receiving palliative care or immediate plans for withdrawal of life sustaining therapy at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional Wall Motion Abnormalities | At the end of delivery of cool blood during continuous dialysis; 12 to 24 hours
  Number of segments undergoing a 20% reduction in longitudinal systolic strain

SECONDARY OUTCOMES:
Regional Wall Motion Abnormalities at 7 days | Seven days after the start of cool blood delivery during continuous dialysis
  Number of segments undergoing a 20% reduction in longitudinal systolic strain after delivery of cool blood during continuous dialysis
Regional Wall Motion Abnormalities at ICU discharge | At ICU discharge, an average of 60 days after the start of cool blood delivery during continuous dialysis
  Number of segments undergoing a 20% reduction in longitudinal systolic strain at ICU discharge
Duration of Continuous Renal Replacement Therapy (CRRT) | Through study completion, an average of 60 days
  Number of hours of CRRT therapy during ICU admission
Renal Recovery at 7 days after cool blood continuous dialysis requiring acute kidney injury | Seven days after the start of cool blood delivery during continuous dialysis
  Renal recovery may best be defined as a reduction in AKI stage at seven days after the start of cool blood continuous dialysis treatment determined by creatinine level and urine output.
Renal Recovery at 24 hours after cool blood continuous dialysis requiring acute kidney injury | 24 hours after the start of cool blood delivery during continuous dialysis
  Renal recovery may best be defined as a reduction in AKI stage at 24 hours after the start of cool blood continuous dialysis treatment determined by creatinine level and urine output.
Low blood pressure | Through study completion, an average of 60 days
  Systolic blood pressure less than 90mmHg or more than 20mmHg fall below baseline; 10% increase in vasopressor dose leading to an increase in blood pressure.
Cumulative vasopressor dose | Through study completion, an average of 60 days
  Dose of vasopressor drugs - unit dependent on drug
Patient's Core Body Temperature (Celsius degrees) | Through study completion, an average of 60 days
  Core body temperature as measured with SpotOn device
Temperature of venous blood in return line (Celsius degrees) | Through study completion, an average of 60 days
  Blood temperature measured with SpotOn device
Intensive care unit free days | After an average of 60 days in the ICU
  Number of days that a participant has been discharged from the ICU while admitted to the hospital
ICU length of stay | Through study completion, an average of 60 days
  Number of days a participant stayed in the ICU
Hospital length of stay | Through study completion, an average of 60 days to hospital discharge
  Number of days a participant stayed in the hospital
ICU mortality | Through study completion, an average of 60 days
  Mortality rate during ICU admission
In Hospital Mortality | Through study completion, an average of 60 days to hospital discharge
  Mortality rate during in hospital stay
60-day Mortality | From study start to up to 60 days from study start
  Mortality rate within the 60 day period
Temperature correlation between nasopharyngeal, forehead, and oral temperature measurements | From study start to up to 60 days from study start
  To correlate invasive measurements of core body temperature (nasopharyngeal) with non-invasive oral and forehead temperature monitoring using the SpotOn system

CONTACTS AND LOCATIONS:
Overall Officials: Marat Slessarev, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Critical Care Trauma Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No